CLINICAL TRIAL: NCT01614951
Title: Pulmonary Dysfunction After Open Heart Surgery: Randomized Clinical Trial With Focus on Lung-protective Interventions
Brief Title: The Pulmonary Protection Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Daniel Steinbruchel, Prof. dr. med., Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4141; 2011-006290-25 (EudraCT Number); 4141 (Other: EudraCT Protocol kode); H-1-2012-0 24 (Other: The Danish Scientific Ethical Committee protocol code); 2007-58-0015. (Other: The Danish Data Protection Agency journal number)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Bretschneider cardioplegic solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pulmonary perfusion (Experimental)
  Interventions: Procedure: Perfusion of the lungs
- Pulmoplegia (Experimental)
  Interventions: Drug: HTK Custodiol
- Control group (Other)
  Interventions: Other: Standard ECC

INTERVENTIONS:
Procedure: Perfusion of the lungs — Pulmonary perfusion with oxygenated blood during ECC.
  Arms: Pulmonary perfusion
Drug: HTK Custodiol — Pulmoplegia before ECC.
  Arms: Pulmoplegia
Other: Standard ECC — ECC after standard procedure
  Arms: Control group

SUMMARY:
The purpose of this study is to investigate whether patients with a preoperative reduced pulmonary function have a better preserved oxygenation capacity after open heart surgery, using either pulmonary perfusion or pulmoplegia compared with TAVI and the control-group with standard ECC (Extra Corporal Circulation).

ELIGIBILITY:
Inclusion Criteria:

1. Planned and urgent surgery on legally competent patients over 18 years:

   * Coronary Artery Bypass Graft Surgery
   * Aortic Valve Replacement
   * Coronary Artery Bypass Graft Surgery + Aortic Valve Replacement
   * Transcatheter Aortic-Valve Implantation
2. Spirometry FEV1 measurement show less than or equal to 80% of the anticipated. We expect that these patients provide the largest signal with lung protective interventions in relation to lung healthy patients.

Exclusion Criteria:

* Previous surgery on the heart or lungs
* Previous thoracic irradiation
* Preoperative heart failure (ejection fraction below 20%).
* Surgical demanding mitral regurgitation
* Unstable patients (heart rate above 100 and systolic blood pressure below 100 mmHg)
* Intubated patients
* Patients with an ongoing preoperative treatment with antibiotics for suspected pneumonia.
* Patients with renal insufficiency requiring hemodialysis
* Pregnant and lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Oxygenation Index | From pre operation until 24 hours post operation
  To investigate whether patients with a preoperative reduced pulmonary function have a better preserved oxygenation index after open heart surgery, using either pulmonary perfusion or pulmoplegia compared with TAVI and the control-group with standard ECC (Extra Corporal Circulation).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A. Steinbrüchel, prof., Principal Investigator — Rigshospitalet, Thoracic Surgery
Locations (1):
- Rigshospitalet, Copenhagen N, Denmark

REFERENCES:
- [Derived] Risom EC, Buggeskov KB, Mogensen UB, Sundskard M, Mortensen J, Ravn HB. Preoperative pulmonary function in all comers for cardiac surgery predicts mortalitydagger. Interact Cardiovasc Thorac Surg. 2019 Aug 1;29(2):244-251. doi: 10.1093/icvts/ivz049. Epub 2019 Mar 15. PMID 30879046
- [Derived] Buggeskov KB, Sundskard MM, Jonassen T, Andersen LW, Secher NH, Ravn HB, Steinbruchel DA, Jakobsen JC, Wetterslev J. Pulmonary artery perfusion versus no pulmonary perfusion during cardiopulmonary bypass in patients with COPD: a randomised clinical trial. BMJ Open Respir Res. 2016 Sep 6;3(1):e000146. doi: 10.1136/bmjresp-2016-000146. eCollection 2016. PMID 27651908
- [Derived] Buggeskov KB, Jakobsen JC, Secher NH, Jonassen T, Andersen LW, Steinbruchel DA, Wetterslev J. Detailed statistical analysis plan for the pulmonary protection trial. Trials. 2014 Dec 23;15:510. doi: 10.1186/1745-6215-15-510. PMID 25539792
- [Derived] Buggeskov KB, Wetterslev J, Secher NH, Andersen LW, Jonassen T, Steinbruchel DA. Pulmonary perfusion with oxygenated blood or custodiol HTK solution during cardiac surgery for postoperative pulmonary function in COPD patients: a trial protocol for the randomized, clinical, parallel group, assessor and data analyst blinded Pulmonary Protection Trial. Trials. 2013 Jan 31;14:30. doi: 10.1186/1745-6215-14-30. PMID 23363494